CLINICAL TRIAL: NCT02769793
Title: Efficacy of Levodopa/Benserazide Dispersible Tablet on Response Fluctuations in Parkinson's Disease Patients With Delayed ON: a Multicenter Randomized Open-label Cross-over Trial
Brief Title: Efficacy of Levodopa/Benserazide Dispersible Tablet on Response Fluctuations in PD Patients With Delayed ON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jee-Young Lee, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-2015-52
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; benserazide, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levodopa dispersible (Experimental): Levodopa dispersible 100mg/tablet, PO, 1 tablet in the morning, once daily for 4 weeks (crossover)
  Interventions: Drug: Levodopa dispersible
- Levodopa (Active Comparator): Levodopa 100mg/tablet, PO, 1 tablet in the morning, once daily for 4 weeks (crossover)
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa dispersible — Levodopa dispersible 100mg/tablet, PO, 1 tablet in the morning, once daily for 4 weeks (crossover)
  Other Names: Madopar dispersible
  Arms: Levodopa dispersible
Drug: Levodopa — Levodopa 100mg/tablet, PO, 1 tablet in the morning, once daily for 4 weeks (crossover)
  Other Names: Madopar
  Arms: Levodopa

SUMMARY:
The purpose of this study is to determine whether levodopa/benserazide dispersible is effective in the adjunctive treatment of Parkinson's disease (PD) patients with delayed ON.

DETAILED DESCRIPTION:
Delayed ON is one of the motor complications of advanced PD patients that effect of anti-parkinsonian medication is delayed more than 40 minutes after intake. In the most severe cases, the effect does not appear even until next medication schedule, so called "No ON" status. It is important to manage delayed ON properly because it can interfere motor functions and quality of life of PD patients.

Levodopa/benserazide dispersible can be absorbed rapidly in the intestine, so theoretically it can break the poor response to conventional treatment of PD patients with delayed ON. However, this has not been proven by clinical trials till now.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 31 and 80 years
* Parkinson disease (PD) was diagnosed by United Kingdom Parkinson disease brain bank criteria
* Patients receiving stable Levodopa treatment at least 2 weeks prior to baseline visit
* Delayed ON was confirmed by a specialized PD diary that records change in motor symptoms 90 minute after the first morning dose. Delayed ON is defined as delay of more than 40 minutes after the first morning dose for resolution of OFF state or experience of no ON state at least 1 per week.

Exclusion Criteria:

* Existence of cognitive decline hard to participate in the clinical trial or K-Minimental Status Exam score 24 or less
* Any contraindication of blood sampling
* Subjects with clinically significant psychiatric illness
* Subjects with a cancer or severe medical illness
* Lactating, pregnant, or possible pregnant
* History of malignant melanoma
* Subjects with narrow-angle glaucoma
* Subjects with hypersensitivity to levodopa or benserazide
* Subjects treated with non-selective monoamine oxidase (MAO)-B inhibitors
* Subjects with peptic ulcer, colitis, or gastrointestinal disease

Ages: 31 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in the time to ON after first morning dose using 3-day PD diary | 4 weeks
  A specialized 3-day PD diary will be distributed to the patients 3 days prior to each visit. This diary will evaluate the latency of ON after intake of the study medication.

SECONDARY OUTCOMES:
Change in the The Unified Parkinson Disease Rating Scale (UPDRS) | 4 weeks
  a scale for assessment of parkinsonian symptom severity in PD patients
Change in the The Unified Dyskinesia Rating Scale (UDyskRS) | 4 weeks
  a scale for assessment of levodopa-induced dyskinesia in PD patients
Change in the The Schwab & England Activity of daily living scale (SEADL) | 4 weeks
  a scale for activity of daily living assessment
Change in the The Parkinson Disease Questionnaire-39 (PDQ-39) | 4 weeks
  a scale for health-related quality of life in PD patients
Change in the Patient global improvement (PGI) | 4 weeks
  patient-centered assessment of global improvement
Change in the Clinician global improvement (CGI) | 4 weeks
  clinician's assessment for global improvement
Change in the K-Minimental status examination (K-MMSE) | 4 weeks
  global cognition assessment
Change in the Total ON time, total OFF time using 3-day PD diary | 4 weeks
  a severity assessment index for PD patients with motor fluctuation

OTHER OUTCOMES:
relationship between delayed ON and response to investigational drugs and the Helicobactor pylori serology and index for atrophic gastritis | at baseline and after 4 weeks of each treatment arm
  whether delayed ON and treatment response are affected by H.pylori status

CONTACTS AND LOCATIONS:
Overall Officials: Jee-Young Lee, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No